CLINICAL TRIAL: NCT07234331
Title: Multicentre Study Analysing Wastewater to Monitor Bacterial Resistance to Antibiotics in Residential Care Homes for Elderly Dependents
Acronym: E-FLUENT
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0586
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Antimicrobial Resistance
Keywords: Nursing home; Wastewater; Surveillance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to model the relationship between the prevalence of ESBL-E and CPE carriage among nursing home residents and their respective concentrations in wastewater discharged from the facility.

DETAILED DESCRIPTION:
Extended-spectrum beta-lactamase-producing Enterobacterales (ESBL-PE) are now endemic in France, complicating the management of infections. In parallel, carbapenemase-producing Enterobacterales (CPE) are exhibiting rapid growth, necessitating enhanced surveillance systems and preventive measures across the healthcare network.

Current antimicrobial resistance (AMR) surveillance systems, which rely primarily on clinical samples, underestimate the dissemination of commensal bacteria and therefore limit the ability to anticipate epidemic events.

Transmission of ESBL-PE and CPE has been documented in long-term care facilities (LTCFs), where they may play a significant role in amplifying and maintaining outbreaks within the healthcare network. However, no dedicated surveillance system currently exists in these facilities.

The current French national strategy is based on standard precautions, but improved detection and identification of ESBL-PE and CPE in LTCFs could enable more effective prevention of transmission and reduce control-related costs.

The primary objective of this study is to model the relationship between the prevalence of ESBL-PE and CPE carriage among LTCF residents and their respective concentrations in facility wastewater effluents.

The primary outcome measure will be the fit and predictive performance of the model for estimating the prevalence of ESBL-PE/CPE carriage among LTCF residents. Carriage prevalence will be assessed through stool sampling or, when unavailable, rectal swabbing. The explanatory variable will be the quantification of ESBL-PE/CPE or resistance genes in wastewater effluents discharged from the LTCF during the corresponding study period.

ELIGIBILITY:
Inclusion Criteria:

* Residents present on the day of sampling (D0 or D+1) in a facility selected during randomization, without criteria regarding length of stay in the facility, and whose health status on the day of the survey permits it;
* Residents who, based on clinical criteria (including an MMSE greater than or equal to 20), are deemed by the nursing home team to be able to understand the issues of the study and to express an informed non-opposition; OR Residents who the nursing home team considers unable to express an informed non-objection but who have a legal representative, a trusted person, or a loved one capable of understanding the information and expressing an informed non-objection.

Residents may be included regardless of the presence of infection, diarrheal stools, antibiotic use or any other treatment, or health status.

Participants in this study may participate in other research projects concurrently.

Exclusion Criteria: Health and medico-social facilities not considered nursing homes (e.g., FAM, MAS, etc.);

* Residents whose health status is incompatible with performing the procedure on the day of the survey (e.g., end-of-life with comfort care);
* Residents with a Mini Mental State Examination (MMSE) score of less than or equal to 20, or without an MMSE score but who, according to nursing home professionals, are unable to provide an informed non-objection and who do not have a legal representative, trusted person, or relative capable of receiving information and providing an informed non-objection;
* Residents, regardless of their MMSE score, who refuse to have the sample taken on the day of the survey even if their legal repre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nursing home residents located in Loire-Atlantique and Maine-et-Loire, France
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Predictive performance | 15 months
  The primary endpoint will be the adequacy and predictive performance of the model for estimating the prevalence of ESBL-E/CPE carriage among nursing home residents. Carriage prevalence will be measured by collecting stool samples from residents or, failing that, by anorectal swabs.

SECONDARY OUTCOMES:
Epidemiology of ESBL/CPE in nursing homes | 15 months
  To assess the prevalence of residents carrying ESBL and CPE in the population of nursing home residents in Loire-Atlantique and Maine-et-Loire
  * Model the relationship between infected residents, ESBL carriers on the one hand, and CPE on the other, and the concentration in wastewater
  * To analyze the factors associated with the prevalence of EBLSE and CPE

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU d'Angers, Angers
  - CHU de Nantes, Nantes